CLINICAL TRIAL: NCT01969474
Title: Phase 1 Study to Study the Efficacy and Safety of Cannabis in the Treatment of Tinnitus
Brief Title: Effectiveness of Cannabis in the Treatment of Tinnitus Patients
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Oron Yahav, MD, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1.01
Record Dates: First submitted 2013-10-14; First posted 2013-10-25 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Tinnitus
Keywords: Tinnitus Cannabis
MeSH Terms: conditions — Tinnitus | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cannabis (Experimental): Treatment with a Cannabis capsule
  Interventions: Drug: Cannabis
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabis — Cannabis capsules given once daily for a month
  Arms: Cannabis
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The hypothesis of the study is that the use of Cannabis will attenuate the tinnitus level as experienced by the patients.

ELIGIBILITY:
Inclusion Criteria:

* Tinnitus lasting more than 3 months
* Tinnitus Handicap Inventory score over 58
* Treated previously for tinnitus (2 modalities)

Exclusion Criteria:

* Prior use of drugs
* Current use of Cannabis
* Neurologic or Psychiatric disease
* Heart Failure
* Ischemic Heart Disease
* Immune Deficiency
* Acoustic Neuroma

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Tinnitus handicap inventory score | 2 months
  Patients will be monitored during a month (treatment time) and a month later

CONTACTS AND LOCATIONS:
Locations (1):
- Wolfson Medical Centre, Holon, Israel